CLINICAL TRIAL: NCT07296900
Title: International Genetic Obesity Registry
Acronym: iGO Registry
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Julia von Schnurbein, PD Dr. med., University of Ulm
Other Study IDs: iGO Registry
Record Dates: First submitted 2025-11-25; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Genetic Obesity
Keywords: genetic obesity; patient registry; monogenic obesity; natural history

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Genetic obesity results from changes in specific genes that affect appetite regulation, metabolism, and fat storage. Its severity and associated health issues vary depending on the genetic cause. In some cases, hormonal imbalances, developmental delays, or other complications may also occur. Identifying the genetic cause is essential for personalized treatment and understanding potential symptoms.

As genetic obesity is rare, specialists often encounter few patients with diverse genetic backgrounds and clinical features. Therefore, collecting global data is crucial to improve our understanding of the condition's progression, complications, and treatment responses for each genetic subtype.

To support this, the International Genetic Obesity Registry (iGO Registry) has been established to gather detailed patient information on genetic obesity. This registry will help advance research and improve clinical care for affected individuals. It will collect data from routine outpatient visits, focusing on relevant diagnostic and treatment information on an international level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with

  * genetically confirmed genetic obesity (ACMG classification 3-5, associated with obesity) and/or
  * early onset severe obesity (BMI ≥ 120% 95th percentile or ≥ 35 kg/m2 before 5 years of age) if genetic testing was performed
* Capable of understanding the aims of the protocol and to provide informed consent (for children and chronically incapacitated individuals, consent is given by their legal guardians)

Exclusion Criteria:

* Not capable of understanding the aims of the protocol and to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Multi-Center
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2075-11 (Estimated); Study Completion 2075-11 (Estimated)

PRIMARY OUTCOMES:
Change of somatic comorbidities under standard treatment | every 5 years for 50 years
  Number of participants with abnormal physical examination findings under standard treatment. Physical examinations include: Body weight [kg], body height [cm], blood pressure [mmHg], heart rate [bpm].
Change of somatic comorbidities under standard treatment | every 5 years for 50 years
  Number of participants with abnormal laboratory test results. Laboratory measurements include. HbA1c [%], blood lipids [mmol/l], insulin [mU/l], glucose [mg/dl]

SECONDARY OUTCOMES:
genotype-phenotype correlation | every 5 years for 50 years
  molecular genetic results will be compared to results from standardized physical examination, laboratory and instrument based tests
Age at onset for comorbidities | every 5 years for 50 years
  comorbidities will be assessed via standard physical examination, laboratory and instrument based tests
Age at death | at year 20 after study start
  patients are followed regulary, age at death (years) will be documented

CONTACTS AND LOCATIONS:
Locations (1):
- Ulm University Clinic, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Yes
Researches participating in the iGO registry and third parties independently can request to perform research with the data.